CLINICAL TRIAL: NCT06215599
Title: Attitude Change Of Hearing Health Professionals On Bone-Anchored Hearing Devices Over Time In a Developing Country
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Head of Dep of Otolaryngology, Pamukkale University
Other Study IDs: 16
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hearing Loss; Bone Anchored Hearing Aids
MeSH Terms: conditions — Hearing Loss | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical doctors: Medical doctors that specialize in ENT and also mostly work in otology
  Interventions: Other: Survey
- audiologist: Health professionals that specialüze in Audiology
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The survey consisted of 14 questions that thoroughly examined the participants' knowledge levels of these conditions, as well as their indication preferences related to BAHIs.

SUMMARY:
This study aims to examine shifts in attitudes about bone-anchored hearing instruments (BAHIs) among hearing health professionals over a period of time.

DETAILED DESCRIPTION:
A survey was designed to assess the knowledge and attitude of participants concerning BAHIs. The survey was administered in both 2019 and 2023 at various conferences, with the questionnaires placed on chairs in different rooms. Responses were collected from Otorhinolaryngologists and audiologists for analysis.

ELIGIBILITY:
Inclusion Criteria:

Working as a licensed health professional as a medical doctor or an audiologist -

Exclusion Criteria:

None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the questionnaire was distributed to participants during relevant congresses of both groups. Consequently, participation was secured from nearly all regions of the country, representing medical institutions at different levels.
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge about BAHI's | Between-2019-2023
  Surveys taht ask about "What is the indicaions of BAHI?" were applied at two time points 2019 and 2023

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)